CLINICAL TRIAL: NCT05299827
Title: Examination of Trunk and Lower Extremity Biomechanics in Children With Lower Urinary System Dysfunction.
Brief Title: Examination of Trunk and Lower Extremity Biomechanics in Children With LUTD.
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Tugtepe Pediatric Urology Clinic (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, Associate professor, Istanbul University - Cerrahpasa
Other Study IDs: IUC-001
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Lower Urinary Tract Symptoms; Posture Disorders in Children; Muscle Weakness Condition; Urinary Incontinence in Children; Lower Extremity Problem
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children diagnosed with lower urinary system dysfunction (LUTD Group): Children who are between the ages of 5-18 and diagnosed with lower urinary system dysfunction by pediatric urologist.
  Interventions: Other: The same evaluation methods were used for both groups.
- Healty Group: Healthy participants in the same age group in the control group; The siblings or cousins of the cases who applied to Tuğtepe Pediatric Urology Center but did not meet the inclusion and exclusion criteria and/or the cases who applied to the outpatient clinic were determined to be healthy after being examined by the relevant physician, and consisted of girls and boys who volunteered to participate in the study. .
  Interventions: Other: The same evaluation methods were used for both groups.

INTERVENTIONS:
Other: The same evaluation methods were used for both groups. — No treatment applied to participants and same evaluation methods used in both groups. Trunk muscle strength, muscle endurance, posture, flexibility and pelvic floor muscle activity of participants was evaluated with stabilizer pressurized biofeedback unit, sit-ups and modified push-ups test; trunk flexors endurance test and Modified Biering Sorensen Test; Posture Screen Mobile And Foot Posture Index; sit-reach-test and Beighton Score; and NeuroTrac-Myoplus4Pro,

SUMMARY:
This study aimed to examine trunk and lower extremity biomechanics among children with lower urinary tract dysfunction (LUTD). It was targeted to pioneer including biomechanical changes into treatment if detected in the trunk and lower extremities of children. Voluntary participants meeting inclusion criteria were divided into two groups: the LUTD group (n=43) and the healthy group (n=43). No treatment was applied to participants and the same evaluation methods were used in both groups. Trunk muscle strength, muscle endurance, posture, flexibility, and pelvic floor muscle activity of participants was evaluated with stabilizer pressurized biofeedback unit, sit-ups and modified push-ups test; trunk flexors endurance test and Modified Biering Sorensen Test; Posture Screen Mobile And Foot Posture Index; sit-reach-test and Beighton Score; and NeuroTrac-Myoplus4Pro, respectively. In addition, the quality of life of participants was evaluated with Pediatric Quality of Life Inventory (PedsQL).

DETAILED DESCRIPTION:
A detailed evaluation is of great importance in the correct diagnosis and treatment of patients with LUTD. In order for a holistic evaluation to show the right path, history taking and physical examination are the most important steps of the evaluation. In addition, it is recommended by ICCS to observe and question the conditions that may cause urgency, holding maneuvers and behavioral structure of the patient. In current clinical practice, changes in posture and balance have been noticed during physiotherapy assessments in children and adolescents with incontinence. In addition, we think that it is possible to disrupt the trunk and lower extremity alignments, which are frequently performed by children with incontinence. These changes may be an important part of the physical and developmental disturbances in children with incontinence. The pelvis and lower extremity consist of interconnected closed chain structures. The movement of any link in the chain depends on the movement and positions of the other links. Therefore, disruption of the alignment of one of the links forming and affecting the chain may cause a change in the mobility and stability of all mechanically related structures, and may also affect the optimal force and activation that the pelvic floor muscles can produce. Our study hypothesizes that the movement of any link in the closed chain of the body and the disruption of one of the links forming this chain cause a change in the mobility, stability and balance of all structures that are mechanically connected, this change will closely affect the activation of the pelvic floor muscles, as well as the children in this group. It was stated that the trunk and lower extremity alignment might have been impaired due to the holding maneuvers that he frequently performed.

Our study, it was aimed to examine the trunk and lower extremity biomechanics in children with LUTD. In addition, if biomechanical changes are detected in the trunk and lower extremities of children and adolescents with incontinence, our study will lead to the necessity of including these changes in the treatment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of the study group (individuals diagnosed with LUTD):

* The cases are between the ages of 5-17
* Having recently been diagnosed with LUTD by a pediatric urologist according to the criteria set by the ICCS
* Not having a diagnosis of enuresis (bedwetting at night) according to the criteria set by ICCS
* Have not received pelvic floor physiotherapy in the last 6 months

Inclusion criteria of the control group (Healthy individuals):

* To be between the ages of 5-17
* Healthy children without LUTD diagnosis and complaints

Exclusion Criteria:

* Having been diagnosed with primary nocturnal enuresis
* Having been diagnosed with neurogenic lower urinary tract dysfunction
* Existence of any condition (cognitive impairment, mental retardation, etc.) that will prevent the parent and child from answering the questions and completing the self-report scales
* Having an orthopedic disease that would prevent evaluation or undergoing surgery that would affect trunk and lower extremity biomechanics
* Presence of anatomical changes and malformations in the urinary system

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants aged 5-18 years who were newly diagnosed with lower urinary tract dysfunction and healthy participants in the same age group.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Deep Trunk Muscle Strength | Baseline
  The measurement of the contraction force of the transversus abdominis from the deep trunk muscles was performed with the Stabilizer Pressure Biofeedback Unit (Chattanooga Stabilizer, USA).Participants were placed in the prone position on a triple inflated object attached to a manometer. Participants were instructed to lie down with the knees straight, spine straight, and head in a comfortable position by placing the inflated object in the lower part of the abdominal region with its long lower edge parallel to the crista iliacas. After the pressure of the manometer was adjusted to 70 mmHg, the participants were asked to slowly contract the transversus abdominis muscle with the abdominal corset technique and maintain this contraction for 5 seconds without holding their breath. Three measurements were recorded and averaged.
Sit-ups Test | Baseline
  With the knees in the flexed position and the feet stabilized, the participants were asked to flex the trunk. During the evaluation, it was recorded how many times the participants were able to perform the movement for 30 seconds.
Modified Push-ups Test | Baseline
  The subjects were positioned prone, knees on the floor, legs flexed, trunk on the floor, elbows flexed, and trunk on the side. From this position, they were asked to raise the head, shoulders and trunk from the ground with the elbows fully extended. During the evaluation, it was recorded how many times the participants were able to do it for 30 seconds.
Trunk Flexors Endurance Test | Baseline
  The participants took positions with the trunk flexed to 60º, knees and hips to 90º flexion. The test was terminated as soon as 60° of trunk flexion was impaired. The time that the participant held this position was recorded in seconds.
Modified "Biering-Sorensen" Test | Baseline
  With this test, the endurance of trunk extensors was evaluated. Participants were positioned in the prone position with the pelvis, hips and knees in full contact with the treatment bed. The participants' pelvis was supported with a belt and fixed by the physiotherapist. The participants were asked to extend their upper body straight forward from the edge of the table, extend it and stay in this position. The time he was able to hold this position properly was recorded in seconds.
Posture Assessment | Baseline
  The postures of the participants were evaluated with the ''Posture Screen Mobile Application''. Front and side photos of the participants were taken with an iOS software phone positioned on a tripod. On the software, the original points determined in the application were marked using the touch screen. According to the reference points, the postural disorder values and the degree of the disorder were calculated for each patient in "cm" via the software and reported. Angular values were expressed as "degrees" (⁰), and distance and offset distances were expressed as "cm". The photographs taken for analysis were digitized using the "Posture Screen" mobile application and the analysis was done through the application.
Foot Posture Index (FPI-6) | Baseline
  For posture analysis of the foot, evaluation was made while the participant was standing and in a relaxed position. Within the scope of FPI-6, bulging in the talonavicular joint area, the structure of the medial longitudinal arch and abduction or adduction of the forefoot with respect to the hindfoot, palpation of the talus head, inclination above and below the lateral malleolus, pronation/supination position of the calcaneus were evaluated. 0 points for neutral foot, positive points for pronation. , a negative score indicates supination. Total scores for left and right feet were recorded separately.
Sit and Reach Test | Baseline
  In order to determine flexibility, the participants were asked to sit on the floor, stretch their legs and rest their soles on a 32 cm high and 35 cm long coffee table without shoes. They were asked to reach forward as far as they could on the coffee table without bending their waist, hips and knees. Participants lie down with their right knee bent, left knee bent, and both knees fully lying on the floor. The distance between the fingers of the distal tip of the middle finger of the hand and the tip of the test table was measured and recorded as cm.
Beighton Score | Baseline
  It is evaluated out of nine points. It is generally accepted that a score of four or more out of nine points indicates hypermobility. In our study, the first four items were evaluated symmetrically in all extremities, as suggested in the scale. Evaluations were made by the participants separately for the movements for the right and left extremities, and 1 point will be given separately for each movement that can be performed on the right-left side. The fifth item includes the whole body. It is the palm touching the ground while standing and knees extended. When this desired movement was performed, it was evaluated as 1 point.

SECONDARY OUTCOMES:
Dysfunctional Voiding and Incontinence Scoring System | Baseline
  Dysfunctional Voiding and Incontinence Scoring System (DVISS) is a 13-item questionnaire. Parents are the target audience. DVISS scores are based on the estimated odds ratio for each question between cases and controls. For example, 1 point is awarded if the odds ratio value is between 2 and 10, and 5 points if it is greater than 50. The total score can range from 0 to 35. A cut-off value of 8.5 shows 90% specificity and sensitivity in detecting BBD.
Childhood Bladder and Bowel Dysfunction Questionnaire (CBDDQ) | Baseline
  The CBBDQ is a parent-filled questionnaire to assess and quantify symptoms of bladder and bowel dysfunction in pediatric patients. The questionnaire is for children aged 5-12 years who have problems with voiding and defecation. Turkish validity and reliability were determined by Aydın et al. Made by in 2020. The Turkish version of the questionnaire consists of 18 questions. The most important features of the questionnaire are that it is short, can be filled in about 5-10 minutes, and is easy to administer and score. Parents were asked to indicate the presence of symptoms in the last month using a five-point Likert scale by ticking the box 0-4. "0" means "no symptoms", "4" means "symptoms occur almost daily. Symptoms worsen as the total score increases.
Pelvic Floor Muscle Activation Measurement | Baseline
  The pelvic floor physiotherapist positions the participant in the butterfly position with support under the legs while lying on their back. Before EMG evaluation, all participants are taught to perform isolated contraction and relaxation of the pelvic floor muscles without the use of accessory muscles by anus palpation. Two superficial electrodes (30 mm diameter (VS30)) are then placed bilaterally adjacent to the mucocutaneous line of the anus at 2 and 7 o'clock to prevent cross-talking (electrodes interference and artifact formation). The reference surface electrode is placed on the inside of the right thigh.
  After proper placement of the electrodes, pelvic floor muscle activity will be measured with the NeuroTrac Myoplus4 Pro device.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya Mutlu, Assoc. Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Tugtepe Pediatric Urology Center, Istanbul, Turkey (Türkiye)